CLINICAL TRIAL: NCT02244268
Title: Effect of ALNA® (Tamsulosin) on the Primary Symptoms of BPH (Benign Prostatic Hyperplasia) Syndrome
Brief Title: Study to Evaluate the Effect of ALNA® (Tamsulosin) on the Primary Symptoms of Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.20
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patient with symptomatic of benign prostatic hyperplasia
  Interventions: Drug: ALNA®

INTERVENTIONS:
Drug: ALNA®
  Other Names: tamsulosin

SUMMARY:
The aims of this observational study are to identify the primary BPH symptoms responsible for the patients to consult a urologic practice, resulting in the prescription of ALNA®, to assess the clincial efficacy on an improved occupational performance of the patients being still employed. Additionally to obtain relevant information for the 5-year report of experience with this product according to the requirements in § 49, para 6 of the German Medicines Act.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from symptomatic benign prostatic hyperplasia (BPH) symptoms and receiving ALNA® treatment are to be included in the observation according to the prescribing information

Exclusion Criteria:

No exclusion criteria is defined, prescribing information is to be considered

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from symptomatic benign prostatic hyperplasia (BPH) syndrome recruited in urological practices
Sampling Method: Non-Probability Sample
Enrollment: 3629 (Actual)
Dates: Start 2000-10; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Change in obstructive BPH symptoms | up to 12 weeks
Change in irritative BPH symptoms | up to 12 weeks

SECONDARY OUTCOMES:
Change in Residual Urine volume | up to 12 weeks
Number of patients with adverse events | up to 12 weeks
Assessment of the number of days on sick leave | up to 12 weeks
Global assessment of efficacy by investigator on a 4-point scale | after 12 weeks
Change in Quality-of-Life Index | up to 12 weeks
Global assessment of tolerability by investigator on a 4-point scale | after 12 weeks
Changes in urinary flow rate | up to 12 weeks